CLINICAL TRIAL: NCT01371123
Title: Serum Aluminum Concentration of Pediatric Patients Receiving Long-Term Parenteral Nutrition: Is There a Problem in Canada?
Brief Title: Serum Aluminum Concentration of Pediatric Patients Receiving Long-Term Parenteral Nutrition
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Academic & Clinical Specialist, Project Investigator., The Hospital for Sick Children
Other Study IDs: 1000025865
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Aluminum Contamination of Parenteral Nutrition
Keywords: serum aluminum; parenteral nutrition; children
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- On long-term PN
- Never been on TPN

SUMMARY:
The purpose of this study is to determine whether children on long-term parenteral nutrition (>6 weeks) have serum aluminum concentrations that are higher than children (aged and gender matched) that have never received parenteral nutrition.

DETAILED DESCRIPTION:
Aluminum contamination of parenteral nutrition (PN) solutions has been a concern for decades because of its link to metabolic bone disease (MBD) due to it's high aluminum content. Currently in the United States, FDA regulations are in place to protect American patients on PN from the effects of aluminum (AL) toxicity. Despite these regulations, pediatric patients on PN are still receiving higher than recommended AL intakes from PN.

Unlike the United States, there are no regulations governing AL content of or intakes from PN solutions in Canada. Consequently, the investigators are unaware of the AL content of the various PN solutions given to our patients. The investigators (the authors) have observed that a significant number of our patients on long-term PN (Home PN), have MBD. Some of our patients have also had bone fractures. The investigators have also observed alteration in calcium and phosphate concentrations as well as suppressed PTH. In an effort to understand the etiology of the MBD the investigators have measured serum AL concentrations in our patients and have found them to be high; between 900 - 2000 nmol/L compared to 0 to 220 nmol/L reported in healthy adults. This has led us to believe that there is a significant problem of AL contamination in PN solutions in Canada. Because the investigators are unable to obtain information on the AL content of the various PN solutions from the PN suppliers, the investigators have decided to report on the serum AL concentrations of our patients as well as the AL concentration of a random sample of PN solutions provided to patients. Plasma aluminum concentrations have already been analyzed in each of the cases. Blood was drawn for routine clinical monitoring on each subject after they had been on PN for six weeks or more.

This is the first step towards raising awareness of the potential problem. It is our hope that this will provide initial evidence to help guide Health Canada's decision regarding regulations on AL content in PN solutions in Canada.

ELIGIBILITY:
Inclusion Criteria:

For Cases on Long-term PN:

1. On PN for ≥ 6 consecutive weeks
2. Has had serum AL concentration drawn and recorded in the past

For Control Subjects:

1. Currently patients at the Hospital for Sick Children being followed on an inpatient ward or in an ambulatory clinic
2. Are not on PN and have never received PN in the past
3. Fed by mouth or enterally with feeding tube

Exclusion Criteria:

For Cases on Long-term PN

1. Patients who are on PN for shorter than 6 weeks
2. Patients who never had serum AL concentration measured
3. Patients who received albumin infusion before blood draw for Al concentration
4. Patients on hemodialysis

For Control Subjects

1. Patients who are not able to be matched to a case/subject on long-term PN for age and gender
2. Patients who do not require blood work as a part of routine clinical monitoring
3. Patients who are on PN
4. Patients with known renal impairment
5. Patients who received albumin infusion before blood draw for Al concentration -

Ages: 6 Weeks to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients followed in the Home-TPN program at the Hospital for Sick Children
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
serum aluminum concentration | 5 months
  A 4 ml blood sample will be obtained from each control subject when they are giving blood for routine clinbical purposes. These subjects will be recruited from in-patient wards or ambulatory clinics. The aluminum content of samples (plasma aluminum concentration) will be determined by high resolution sector field inductively coupled mass spectrometry (HR-SF-ICP-MS). The accuracy and precision of the instrument used to determine aluminum concentration is measured using external and internal standards. Accuracy and precision was last measured at ± 0.5 to 2.5% and 5 to 10% respectively

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, MSc, PhD, RD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Courtney-Martin G, Kosar C, Campbell A, Avitzur Y, Wales PW, Steinberg K, Harrison D, Chambers K. Plasma Aluminum Concentrations in Pediatric Patients Receiving Long-Term Parenteral Nutrition. JPEN J Parenter Enteral Nutr. 2015 Jul;39(5):578-85. doi: 10.1177/0148607114531046. Epub 2014 Apr 17. PMID 24743391